CLINICAL TRIAL: NCT02227771
Title: CONventional Antegrade vs Sub-Intimal Synergy sTENTing in Chronic Total Occlusions
Brief Title: Consistent CTO Trial
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Cardiovascular Research Center (Network)
Collaborators: Ceric Sàrl (Industry)
Responsible Party: Sponsor
Other Study IDs: BSC-03
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Chronic Total Occlusion
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patient with chronic total occlusion
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention

SUMMARY:
The purpose of this study is to demonstrate that enhanced vascular healing with the Synergy stent should minimize the risk of late aneurysm formation and potential clinical complications but not at the cost of enhanced efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient >18 years old
* Females of childbearing potential with a negative pregnancy test
* Presence of Chronic Total Occlusion (CTO) that is known or presumed to be of at least 3 months in duration
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent
* Attempt to implant at least one Synergy II stent has been made

Exclusion Criteria:

* Acute myocardial infarction with ongoing ST-elevation
* Cardiogenic shock
* Left ventricular ejection fraction <20%
* Subject has one of the following (as assessed prior to the index procedure):

Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 24 months Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.) Planned procedure that may cause non-compliance with the protocol or confound data interpretation

* Subject is treated by dialysis or has a baseline serum creatinine level >220 μmol/L (2.5 mg/dL)
* Known allergy to to contrast (that cannot be adequately premedicated) and/or the trial stent system or protocol-required concomitant medications (e.g., platinum, platinum-chromium alloy, stainless steel, everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors, or aspirin)
* Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint OR subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* Need for ongoing long-term anticoagulation
* Subject has received an organ transplant or is on a waiting list for an organ transplant
* Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Planned CABG after the index procedure
* Subject previously treated at any time with intravascular brachytherapy
* Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Subject has a white blood cell (WBC) count < 3,000 cells/mm3
* Subject has documented or suspected liver disease, including laboratory evidence of hepatitis
* Subject has a clinically significant bleeding diathesis or coagulopathy or will refuse blood transfusions
* Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
* Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
* Subject has severe symptomatic heart failure (i.e., NYHA class IV)
* Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)
* Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who come to hospital for CTO and who met all the inclusion/eclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 215 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12-31 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The primary stent endpoint is 12-month target vessel failure (TVF) rate | 12 months
  The primary stent endpoint is 12-month target vessel failure (TVF) rate, defined as any ischemia-driven revascularization of the target vessel, MI (Q-wave and non-Q-wave) related to the target vessel or cardiac death.
The primary balloon endpoint is device procedural success | 1 month
  Successful delivery of the Emerge Coronary Dilatation catherter across the lesion and Successful inflation and removal of the Emerge Coronary Dilatation catherter with absences of clinically significant vessel perforation or flow limiting vessel dissection, reduction in thrombolysis in myocardial infarction (TIMI) flow from baseline, clinically significant arrythmias requiring medical treatment or device intervention following dilatation with Emerge balloon and Achievment of final TIMLI 3 flow for the target lesion at the conclusion of the index procedure. The primary balloon endpoint will be evaluated in patients where an attempt to use an Emerge Coronary Dilatation catherter is made.

SECONDARY OUTCOMES:
Target lesion revascularization (TLR) rate | In hospital, 6 Months, 12 Months, 2 Years
Target lesion failure (TLF) rate | In hospital, 6 Months, 12 Months, 2 Years
Target vessel revascularization (TVR) rate | In hospital, 6 Months, 12 Months, 2 Years
Target vessel failure (TVF) rate | In hospital, 6 Months, 12 Months, 2 Years
Myocardial infarction (MI, Q-wave and non-Q-wave) rate | In hospital, 6 Months, 12 Months, 2 Years
Cardiac death rate | In hospital, 6 Months, 12 Months, 2 Years
Non-cardiac death rate | In hospital, 6 Months, 12 Months, 2 Years
All death rate | In hospital, 6 Months, 12 Months, 2 Years
Cardiac death or MI rate | In hospital, 6 Months, 12 Months, 2 Years
All death or MI rate | In hospital, 6 Months, 12 Months, 2 Years
All death/MI/TVR rate | In hospital, 6 Months, 12 Months, 2 Years
Stent thrombosis rate (by ARC definitions) | In hospital, 6 Months, 12 Months, 2 Years
Angina, dyspnoea and quality of life scores | 12 Months
In-stent and in-segment percent diameter stenosis (%DS) | Peri-procedural
In-stent and in-segment minimum lumen diameter (MLD) | Peri-procedural
Acute gain | Peri-procedural
In-stent and in-segment %DS | 12-Months Post-Index Procedure
In-segment late loss | 12-Months Post-Index Procedure
In-stent and in-segment binary restenosis rate | 12-Months Post-Index Procedure
In-stent and in-segment MLD | 12-Months Post-Index Procedure
Incomplete apposition | Peri-procedural
Stent, vessel and lumen areas and volumes | Peri-procedural
Incomplete apposition | 12-Months Post-Index Procedure
Aneurysm formation | 12-Months Post-Index Procedure
Endothelial strut coverage percentage | 12-Months Post-Index Procedure

CONTACTS AND LOCATIONS:
Locations (6):
- United Kingdom (6):
  - Belfast Health & Social Care Trust, Belfast
  - Bristol Royal Infirmary, Bristol
  - Edinburgh Royal Infirmary, Edinburgh
  - Golden Jubilee, Glasgow, Glasgow
  - London Chest Hospital,, London
  - Kings College, London, London

REFERENCES:
- [Derived] Walsh SJ, Hanratty CG, McEntegart M, Strange JW, Rigger J, Henriksen PA, Smith EJ, Wilson SJ, Hill JM, Mehmedbegovic Z, Chevalier B, Morice MC, Spratt JC. Intravascular Healing Is Not Affected by Approaches in Contemporary CTO PCI: The CONSISTENT CTO Study. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1448-1457. doi: 10.1016/j.jcin.2020.03.032. PMID 32553333